CLINICAL TRIAL: NCT04780789
Title: Volumetric Analysis of Hepatocellular Carcinoma After Transarterial Chemoembolization and Its Impact on Overall Survival
Brief Title: Volumetric Analysis of Hepatocellular Carcinoma After Transarterial Chemoembolization
Status: Completed | Type: Observational
Sponsor: Brno University Hospital (Other)
Collaborators: Masaryk Memorial Cancer Institute (Other); Masaryk University (Other)
Responsible Party: Principal Investigator, Monika Hajkova, Principal Investigator, Brno University Hospital
Other Study IDs: 01-080616/EK
Record Dates: First submitted 2021-02-17; First posted 2021-03-04 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Hepatocellular Carcinoma; Hepatocellular Carcinoma by BCLC Stage
Keywords: Transarterial Chemoembolization; RECIST; mRECIST; Volumetric analysis
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Transarterial Chemoembolization — A contrast agent (Xenetix350, Guerbet, France) was applied under local anaesthesia via the common femoral artery using a 5F sheath. Selective catheterization of the coeliac trunk and other arteries supplying the liver was then performed under fluoroscopic control. A pathological vascularization pattern was identified and chemoembolization material consisting of DC beads (BTG International Ltd) was injected by the treating angiographist using micro instrumentation. Follow-up CT or MRI was performed after 1-3 TACE sessions according to the extent of the lesion, 3 weeks following the last procedure. Patients with completed treatments were scheduled for an imaging follow-up every 3 months, allowing evaluation of the effect of treatment. In case of a positive response to the treatment another session of TACE was indicated. Chemoembolization sessions were performed as inpatient procedures with the mean hospitalization time of 4 days.
  Other Names: Transarterial Chemoembolization with Drug-Eluting Beads

SUMMARY:
The application of transarterial chemoembolisation (TACE) with drug-eluting beads in patients with hepatocellular carcinoma and its response to the treatment will be observed. The registry has the following objectives:

To assess the response to the treatment by standard methods and volumetric analysis as well as trying to determine any predictive response factors To determinate interobserver variability of the methods.

DETAILED DESCRIPTION:
The patients with hepatocellular carcinoma in stage suitable for treatment by transarterial chemoembolization (TACE) with drug-eluting beads are included in the study. The investigators assess the response to the treatment by standard methods (RECIST, mRECIST) as well as by volumetric analysis. The size of tumor is evaluated on CT/MRI by two investigators prior to first TACE and then on all the check-ups (routinely every three months) until 31 December, 2019 or the patients' death.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of HCC by a radiologist according to the European Association for the Study of the Liver (EASL) criteria or confirmed histologically
* at least one TACE undergone at the University Hospital Brno
* initial/ closing CT (Brillance 64, Philips, Netherlands; contrast enhancement 125 mL Iomeron 400, Bracco, Germany) or MRI study (Achieva, Philips, Netherlands, SENSE XL Torso coil 16 1.5T; contrast enhancement 15 mL Primovist, Bayer, Germany)
* follow-up on or before December 31, 2019.

Exclusion Criteria:

* when the inclusion criteria are not met.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hepatocellular carcinoma undergoing transrarterial chemoembolization
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Predictive factors for overall survival and progression-free survival | 4 years 11 months
  RECIST, mRECIST, volumetric analysis
Interobserver variability of the methods used for assessing tumor response to the treatment | 4 years 11 months
  RECIST, mRECIST, volumetric analysis

SECONDARY OUTCOMES:
Time from observation until death due to any cause (or censoring) | 4 years 11 months
  Overall survival
Time from observation until disease progression or death | 4 years 11 months
  Progression-free survival
Response to the treatment, as assessed by RECIST (v.1.1) | 4 years 11 months
  Objective Tumour Response will be assessed by the investigators on CT/MRI image analysis
Response to the treatment, as assessed by mRECIST | 4 years 11 months
  Objective Tumour Response will be assessed by the investigators on CT/MRI image analysis
Response to the treatment, as assessed by volumetric analysis | 4 years 11 months
  Objective Tumour Response will be assessed by the investigators on CT/MRI image